CLINICAL TRIAL: NCT06539975
Title: Effectiveness of Evening Primrose Oil for Induction of Labor
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, sayed mohamed sayed mostafa, sayed mohamed sayed mostafa, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: primrose oil in labor
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Induction of Labor
MeSH Terms: interventions — evening primrose oil

STUDY DESIGN:
Intervention Model Description: The study will be a douple-centered, serially-numbered closed opaque envelope, randomised clinical trial.
Who Masked: Investigator
Masking Description: Allocation concealment is the use of sequentially numbered,opaque,sealed envelopes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evening primrose oil + misoprostol (Active Comparator): combination of both drugs for induction of labor adminstrated vaginally.
  Interventions: Drug: Evening Primrose Oil 1000 MG
- misoprostol only (Other): misoprostol alone for induction of labor adminstrated vaginally.
  Interventions: Drug: Evening Primrose Oil 1000 MG

INTERVENTIONS:
Drug: Evening Primrose Oil 1000 MG — Evening primrose oil 1000mg vaginally plus misoprostal for induction of labor

SUMMARY:
Effectivness of primrose oil in induction of labour .

DETAILED DESCRIPTION:
Using primrose oil in addition to misoprostol for induction of labor in one group of pregnant women and compare the result with those of another group in which we are using misoprstol only.

ELIGIBILITY:
Inclusion Criteria:

* pregenent of 38 weeks and longer
* singleton pregenency
* vertex presentation
* indication of labor induction
* bishop score <6 and cervical dilation<2 cm

Exclusion Criteria:

* women who delivered by classical cs or had a history of myomectomy , hysterscopic uterine surgery , or cervical surgery like conisation
* women with multiple gestation
* women with evidence of low implanted placenta by ultrasound
* women with contraindication to misoprostol or vaginal delivery

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 72 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
The interval between induction of labor and delivery | induction of labor may take more than 24 hours
  comparing between the interval between induction of labor and delivery in two groups one is using evening primrose oil + misoprostol and the other using misoprostol only.

REFERENCES:
- [Background] Hemmatzadeh S, Mohammad Alizadeh Charandabi S, Veisy A, Mirghafourvand M. Evening primrose oil for cervical ripening in term pregnancies: a systematic review and meta-analysis. J Complement Integr Med. 2021 Jul 14;20(2):328-337. doi: 10.1515/jcim-2020-0314. eCollection 2023 Jun 1. PMID 34261202
- [Result] Moradi M, Niazi A, Heydarian Miri H, Lopez V. The effect of evening primrose oil on labor induction and cervical ripening: A systematic review and meta-analysis. Phytother Res. 2021 Oct;35(10):5374-5383. doi: 10.1002/ptr.7147. Epub 2021 Apr 29. PMID 33913585